CLINICAL TRIAL: NCT01041313
Title: Memantine for Post-Operative Pain Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Gregory Terman, MD, PhD, Professor, University of Washington, Department of Anesthesiology and Pain Medicine, Division of Pain Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35063-A; NAM-MD-63
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Pain, Post-operative
Keywords: Adjuvants, pharmaceuticals; Receptors, N-Methyl-D-Aspartate; Drug tolerance; Pain Measurement
MeSH Terms: conditions — Pain, Postoperative | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opiate Naive (Active Comparator): Subjects who have not taken opiate medication in previous 6 weeks before surgery
  Interventions: Drug: Memantine; Drug: Placebo
- Opiate tolerant (Active Comparator): Subjects who have taken opiate medications for the 6 weeks before surgery
  Interventions: Drug: Memantine; Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 7 days prior to surgery, start taking 5mg memantine daily; 4 days prior to surgery, increase dose to 5mg twice daily; 2 days prior to surgery, increase dose to 10mg in the morning, and 5 mg in the evening; on the day of surgery, increase dose to 10mg twice daily, and continue on this dose until 14 days after surgery.
  Other Names: Namenda
Drug: Placebo — 7 days prior to surgery, start taking one placebo tablet daily; 4 days prior to surgery, increase dose to one placebo tablet twice daily; 2 days prior to surgery, increase dose to 2 placebo tablets in the morning, and one placebo tablet in the evening; on the day of surgery, increase dose to 2 placebo tablets in the morning and 1 placebo tablet in the evening. On the first day after surgery through 14 days after surgery, take 1 placebo tablet twice daily.

SUMMARY:
Pain is a common element of surgery. Opiates (morphine, oxycodone, hydrocodone, methadone, fentanyl) are very helpful in decreasing pain after surgery. Unfortunately, with repeated use opiates lose their effectiveness, such that patients need to utilize more opiates to achieve adequate pain relief - a phenomenon called tolerance. Sometimes tolerance to a pain reliever's effects can develop in just a few hours. It is thought that activation of the N-methyl d-aspartate (NMDA) receptor, a "switch" found on the surface of nerves, is partially responsible for opiate tolerance. Memantine is a medication that limits the activity of NMDA receptors in the brain and spinal cord. It has been used for years to help patients with Alzheimer's Disease. In this study, we will study the effects of memantine when combined with opiate medications to see whether it can increase the effectiveness of opiates for pain after surgery and reduce the side effects caused by opiates (e.g., sedation, nausea, itching).

ELIGIBILITY:
Inclusion Criteria:

* Surgery for total hip replacement, knee replacement OR lumbar spinal fusion
* Taking no opiate medication OR taking opiate medication for at least 6 weeks

Exclusion Criteria:

* History of alcohol or drug abuse
* Clinical diagnosis of Alzheimer's Disease
* Prior adverse reaction to memantine
* Severe renal impairment (creatinine clearance <30 ml/min)
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Change in numerical ratings on pain diaries as outpatients (pre and post surgery) | For 1 week pre-surgery, through 2 weeks post-surgery
Daily pain numerical ratings at rest and with movement as inpatients. | Immediately post-surgery until discharge (2-3 days)
Total opiate dose via patient controlled IV hydromorphone | Post-surgery day 1
Oxycodone dose taken prn | Post-surgery day 2 through 3 months.

SECONDARY OUTCOMES:
Treatment group differences in side effects (nausea, itching, sedation, urinary retention following foley catheter discontinuation) | One week pre-surgery through 3 months post-surgery
Changes in cognitive function, assessed with Digit-Symbol Substitution Test and Trail Making Test B | One week pre-surgery, immediately pre-surgery, and post-surgery days 1, 2, 3
Changes in pain and quality of life questionnaire responses (SF-McGill-2, Brief Pain Questionnaire, SF-36 v2) | One week pre-surgery through 3 months post-surgery, particularly as outpatient

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Terman, MD, PhD, Principal Investigator — University of Washington Department of Anesthesiology and Pain Medicine
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Grande LA, O'Donnell BR, Fitzgibbon DR, Terman GW. Ultra-low dose ketamine and memantine treatment for pain in an opioid-tolerant oncology patient. Anesth Analg. 2008 Oct;107(4):1380-3. doi: 10.1213/ane.0b013e3181733ddd. PMID 18806055